Statistical analysis

For testing the study hypotheses, the following statistical methods will be used:

- 1. Descriptive statistics (mean and standard deviation) of the demographic data of all patients in both groups.
- 2. The suitable statistical tests will be used according to the nature of the collected data.
- 3. Level of significance for all tests will be set at p-value  $\leq 0.05$ .
- 4. The statistical package for social sciences (SPSS) version 26 for windows (Armonk, NY: IBM Corp) will be used for data statistical analysis.